CLINICAL TRIAL: NCT04991337
Title: Effects of Detraining in Endurance Athletes With Atrial Fibrillation (NEXAF Detraining)
Brief Title: Effects of Detraining in Endurance Athletes With Atrial Fibrillation
Acronym: NEXAF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: St. Olavs Hospital (Other); Baker Heart and Diabetes Institute (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Hospital, Antwerp (Other); AZ Jan Palfijn Gent (Other); Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEXAF Detraining
Record Dates: First submitted 2021-05-07; First posted 2021-08-05 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Atrial Fibrillation
Keywords: heart
MeSH Terms: conditions — Atrial Fibrillation | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two-arm international multicenter open-label randomized (1:1) controlled trial with blinded end-point evaluation.
Who Masked: Outcomes Assessor
Masking Description: Open label study and participants are not blinded to group allocation. Researchers and staff are unblinded during all procedures. AF burden will be adjudicated by a blinded endpoint committee and researchers will be blinded to group allocation when performing statistical analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Detraining group (Experimental): Will be instructed to avoid high-intensity exercise corresponding to a heart rate >75% of maximum heart rate, and a total duration of exercise (hours/week) corresponding to >80% of the self-reported average weekly amount of exercise (hours/week) during the past six months, for a period of 16 week.
  Interventions: Behavioral: Detraining group
- Control group (Experimental): Will be instructed to perform at least three weekly sessions of high intensity exercise, corresponding to a HR ≥85% of maximum heart rate, and otherwise continue endurance exercise as usual.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Detraining group — Detraining is defined as exercise corresponding to a heart rate ≤75% of maximum heart rate and ≤80% of the self-reported average weekly amount of exercise (hours/week) during the past six months, for a period of 16 weeks.
  Arms: Detraining group
Behavioral: Control group — At least three weekly sessions of high intensity exercise, corresponding to a heart rate ≥85% of maximum heart rate, and otherwise continue endurance exercise as usual.
  Arms: Control group

SUMMARY:
Atrial fibrillation (AF) affects more than 43 million people worldwide, but specific exercise recommendations do not exist for this group of patients. Despite a lack of evidence, athletes are often advised to reduce exercise intensity (detraining) after being diagnosed with AF. This randomized controlled trial will be the first study that investigates effects of detraining in endurance athletes. Participants will be randomized to an intervention group that will be instructed to refrain from high intensity exercise, and a control group. The study aims to clarify whether detraining might reduce the burden of AF and has the potential to guide development of exercise guidelines for AF patients.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) affects more than 43 million people worldwide, but specific exercise recommendations do not exist for this group of patients. Despite a lack of evidence, athletes are often advised to reduce exercise intensity (detraining) after being diagnosed with AF. This randomized controlled trial will be the first study that investigates effects of detraining in endurance athletes. Participants will be included at Bærum Hospital, St.Olavs Hospital, Trondheim, Baker Institute, Melbourne, Leuven University Hospital, Antwerp University Hospital, AZ Jan Palfijn Gent and Jessa Hospital Hasselt, Belgium. In total 120 participants will be monitored with a chest-strap heart rate (HR) monitor and sportswatch (exercise intensity), and an Insertable Cardiac Monitor (ICM, AF burden). Participants will be randomized to an intervention group (n=60) that will be instructed to refrain from high intensity exercise (H) >75% of maximal HR (HRmax)) for a period of 16 Weeks, or a control group (n=60) that will be instructed to perform at least three weekly sessions of high intensity training (HR ≥85% of HRmax. The primary endpoint will be AF burden, as measured by continuous monitoring with ICMs and calculated as the cumulative duration of all AF episodes lasting ≥30sec divided by total duration of monitoring. The study aims to clarify whether detraining might reduce the burden of AF and has the potential to guide development of exercise guidelines for AF patients. The investigators will also study exercise-induced cardiac remodeling, aiming to improve the understanding of underlying pathophysiological mechanisms for AF.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* Diagnosed with paroxysmal atrial fibrillation (verified by electrocardiogram)
* Report >5 (running, rowing) or >8 (cycling, cross-country skiing), weekly hours, respectively, of endurance sport
* At least two anamnestic (self-reported) episodes of atrial fibrillation, of which one during the last six months
* Use a smartphone and agree to connect their sportswatch with a web-based platform for monitoring of exercise

Exclusion Criteria:

* Permanent atrial fibrillation
* Cardiac conditions (including valvular heart disease of moderate or greater severity, symptomatic ischemic heart disease)
* Left ventricular ejection fraction <45%
* Hypertension (>140/90)
* Diabetes mellitus
* Hyperthyroidism
* Smoking during the last 5 years
* Alcohol intake >20 alcohol units/week
* Use of illegal or performance enhancing drugs
* Body mass index >30kg/m2
* Injuries preventing physical exercise
* Pregnancy
* Participation in conflicting intervention research studies
* Planned atrial fibrillation ablation within the next six months
* The individual refuses to have an insertable cardiac monitor, blood samples taken or be part of the detraining group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation burden | Measured during the last 4 weeks (week 13-16) of the 16-week intervention period
  Atrial fibrillation burden (time with atrial fibrillation) as measured by continuous monitoring with insertable cardiac monitor and calculated as the cumulative duration of all atrial fibrillation episodes lasting ≥30sec divided by total duration of monitoring and reported as percentages.

SECONDARY OUTCOMES:
Atrial fibrillation burden | Measured during the first 4 weeks (week 1-4) of the 16-week intervention period
  Atrial fibrillation burden as measured by continuous monitoring with insertable cardiac monitor and calculated as the cumulative duration of all atrial fibrillation episodes lasting ≥30sec divided by total duration of monitoring.
Atrial fibrillation burden | Measured during week 5-8 of the 16-week intervention period
  Atrial fibrillation burden as measured by continuous monitoring with insertable cardiac monitor and calculated as the cumulative duration of all atrial fibrillation episodes lasting ≥30sec divided by total duration of monitoring.
Atrial fibrillation burden | Measured during week 9-12 of the 16-week intervention period
  Atrial fibrillation burden as measured by continuous monitoring with insertable cardiac monitor and calculated as the cumulative duration of all atrial fibrillation episodes lasting ≥30sec divided by total duration of monitoring.
Cumulative atrial fibrillation burden | Measured during the entire 16-week intervention period
  Atrial fibrillation burden as measured by continuous monitoring with insertable cardiac monitor and calculated as the cumulative duration of all atrial fibrillation episodes lasting ≥30sec divided by total duration of monitoring.
Atrial fibrillation episode duration | Measured during the 16-week intervention period
  Mean duration of atrial fibrillation episodes lasting ≥30sec
Atrial fibrillation episodes | Measured during the first 4 weeks (week 1-4) of the 16-week intervention period
  Number of atrial fibrillation episodes lasting ≥30sec, as measured by insertable cardiac monitor
Atrial fibrillation episodes | Measured during week 5-8 of the 16-week intervention period
  Number of atrial fibrillation episodes lasting ≥30sec, as measured by insertable cardiac monitor
Atrial fibrillation episodes | Measured during week 9-12 of the 16-week intervention period
  Number of atrial fibrillation episodes lasting ≥30sec, as measured by insertable cardiac monitor
Atrial fibrillation episodes | Measured during the last 4 weeks (week 13-16) of the 16-week intervention period
  Number of atrial fibrillation episodes lasting ≥30sec, as measured by insertable cardiac monitor
Cumulative atrial fibrillation episodes | Measured during the 16-week intervention period
  Number of atrial fibrillation episodes lasting ≥30sec, as measured by insertable cardiac monitor
Days with atrial fibrillation | Measured during the 16-week intervention period
  Days with at least one episode of atrial fibrillation lasting ≥30sec
Days without atrial fibrillation | Measured during the 16-week intervention period
  Days without atrial fibrillation episodes
Relative change in atrial fibrillation burden | Measured during the 4-week baseline period prior to randomization and during the last 4 weeks of the 16-week intervention period
  Relative change in atrial fibrillation burden as measured by continuous monitoring with insertable cardiac monitor and calculated as the cumulative duration of all atrial fibrillation episodes lasting ≥30sec divided by total duration of monitoring
Relative change in atrial fibrillation burden | Measured during the 4-week baseline period prior to randomization and during the first 4 weeks of the 16-week intervention period
  Relative change in atrial fibrillation burden as measured by continuous monitoring with insertable cardiac monitor and calculated as the cumulative duration of all atrial fibrillation episodes lasting ≥30sec divided by total duration of monitoring
Relative change in atrial fibrillation burden | Measured during the 4-week baseline period prior to randomization and during the entire 16-week intervention period
  Relative change in atrial fibrillation burden as measured by continuous monitoring with insertable cardiac monitor and calculated as the cumulative duration of all atrial fibrillation episodes lasting ≥30sec divided by total duration of monitoring
Adherence to prescribed exercise | 16 weeks
  Adherence to prescribed exercise (>80% of exercise with ≥85% and ≤75% of maximum heart rate, respectively)
Exercise capacity | Measured at the baseline study visit and at the final study visit after the 16-week intervention period
  Peak oxygen uptake (VO2peak)
Atrial volumes | Measured at the baseline study visit and at the final study visit after the 16-week intervention period
  Right and left atrial volumes measured with echocardiography
Ventricular volumes | Measured at the baseline study visit and at the final study visit after the 16-week intervention period
  Right and left ventricular volumes measured with echocardiography
Atrial function | Measured at the baseline study visit and at the final study visit after the 16-week intervention period
  Left atrial function measured by strain with echocardiography
Ventricular function | Measured at the baseline study visit and at the final study visit after the 16-week intervention period
  Right and left ventricular function measured by strain with echocardiography
Systolic function | Measured at the baseline study visit and at the final study visit after the 16-week intervention period
  Left ventricular ejection fraction measured by strain with echocardiography
Atrial fibrillation symptoms | Measured by questtionnaire at the baseline study visit and at the final study visit after the 16-week intervention period
  Self-reported number of symptomatic atrial fibrillation episodes
Atrial Fibrillation Effect on QualiTy-of-life questionnaire | Measured at the baseline study visit and at the final study visit after the 16-week intervention period
  Measured with the Atrial Fibrillation Effect on QualiTy-of-life questionnaire (AFEQT).
  Minimum score 0, maximum score 100, higher values indicate better quality of life
Atrial fibrillation hospitalizations | Throughout study completion, an average of 22 weeks
  Number of unplanned hospitalizations due to atrial fibrillation cardioversion or ablation
Modified European Heart Rhythm Association Symptom Scale (mEHRA) symptom classification | Measured at the baseline study visit and at the final study visit after the 16-week intervention period
  Modified European Heart Rhythm Association Symptom Scale (mEHRA) questionnaire. The scale ranges from minimum 1 to maxiumum 4, a higher score indicates a worse symptom burden
Number of ventricular arrhythmias | Throughout study completion, an average of 22 weeks
  Ventricular arrhythmias lasting ≥12 ventricular complexes as measured by continuous monitoring with insertable cardiac monitor
Number of adverse events | Throughout study completion, an average of 22 weeks
  Any unfavorable and unintended sign, symptom or illness that develops or worsens during the trial period will be reported as adverse events (AE). A serious adverse event (SAE) is defined as death, any life-threatening event or any inpatient hospitalisation
Cardiovascular risk factors measured by blood pressure | Measured at baseline and after the 16-week intervention period
  Measure of blood pressure (mmHg)
Cardiovascular risk factors measured by blood lipids | Measured at baseline and after the 16-week intervention period
  Blood lipids (mmol/L)
Cardiovascular risk factors measured by weight | Measured at baseline and after the 16-week intervention period
  Weight (kg)
Cardiovascular risk factors measured by BMI | Measured at baseline and after the 16-week intervention period
  BMI (weight and height will be combined to report BMI in kg/m^2)
Cardiovascular risk factors measured by smoking | Measured at baseline and after the 16-week intervention period
  Smoking (pack years)
Cardiovascular risk factors measured by alcohol units | Measured at baseline and after the 16-week intervention period
  Alcohol use (units)
Cardiovascular biomarkers - inflammation markers | Measured at baseline and after the 16-week intervention period
  Markers for inflammation markers; interleukines and hrCRP (mg/L)
Cardiovascular biomarkers - markers for myocardial damage | Measured at baseline and after the 16-week intervention period
  Markers for myocardial damage, measured by troponin T (ng/L) and NT-ProBNP (ng/L)
Immediate effects on arrhythmia burden of high-intensity exercise | 24 hours after after peak exercise testing
  Ahrrythmias measured with 24-hour electrocardiogram after peak exercise testing
Immediate effects on biomarkers of exercise | At peak exercise during cardiopulmonary exercise testing
  Blood sampling at peak exercise for analyses of cardiac Troponins, NT-pro-BNP, interleukins, C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Marius Myrstad, |MD, PhD, Principal Investigator — Vestre Viken Health trust
Locations (1):
- Vestre Viken Health Trust, Baerum Hospital, Bærums verk, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Apelland T, Letnes JM, Janssens K, Claessen G, Tveit A, Sellevold AB, Mitchell A, Willems R, Onarheim S, Enger S, Kizilkilic SE, Miljoen H, Elliott A, Loennechen JP, La Gerche A, Myrstad M; NEXAF Investigators. Arrhythmia burden, symptoms and quality of life in female and male endurance athletes with paroxysmal atrial fibrillation: a multicentre cohort study in Norway, Australia and Belgium. BMJ Open. 2025 Aug 5;15(8):e100496. doi: 10.1136/bmjopen-2025-100496. PMID 40764068
- [Derived] Apelland T, Sellevold AB, Letnes JM, Onarheim S, Enger S, Tveit A, Delpire B, Claessen G, La Gerche A, Loennechen JP, Berge T, Myrstad M; NEXAF Investigators; NEXAF investigators. Cardiac arrhythmia assessment with patch electrocardiogram versus insertable cardiac monitor: a cohort study in endurance athletes with atrial fibrillation. BMJ Open. 2025 Jan 6;15(1):e093250. doi: 10.1136/bmjopen-2024-093250. PMID 39762092
- [Derived] Apelland T, Janssens K, Loennechen JP, Claessen G, Sorensen E, Mitchell A, Sellevold AB, Enger S, Onarheim S, Letnes JM, Miljoen H, Tveit A, La Gerche A, Myrstad M; NEXAF investigators. Effects of training adaption in endurance athletes with atrial fibrillation: protocol for a multicentre randomised controlled trial. BMJ Open Sport Exerc Med. 2023 Apr 11;9(2):e001541. doi: 10.1136/bmjsem-2023-001541. eCollection 2023. PMID 37073174